CLINICAL TRIAL: NCT05364359
Title: Individuel diætvejledning på Baggrund af Smagstest Hos Patienter Med hæmatologisk Cancer i Cytostatisk Behandling
Brief Title: Individual Dietary Counseling Based on Taste-tests in Patients With Hematological Cancer in Cytostatic Therapy
Acronym: HCP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Copenhagen (Other)
Collaborators: Zealand University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HCP
Record Dates: First submitted 2022-03-23; First posted 2022-05-06 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Hematological Malignancy
Keywords: cancer; hematological; malignancy
MeSH Terms: conditions — Hematologic Neoplasms; Neoplasms | interventions — Nutrition Assessment; Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): The patients will receive a individual dietary counseling based on the taste-test
  Interventions: Dietary Supplement: Taste-test
- Standard dietary counseling (Placebo Comparator): The patients will receive a individual standard dietary counseling not based on the taste-test
  Interventions: Other: Standard care

INTERVENTIONS:
Dietary Supplement: Taste-test — Patients will receive a dietary counseling based on a simple taste-test
  Other Names: Dietary counseling
  Arms: Intervention group
Other: Standard care — Patients will receive a dietary counseling based on a standard dietary counseling for the patient group
  Arms: Standard dietary counseling

SUMMARY:
The purpose of the study is to investigate whether a simple taste-test will increase the intake of energy as part of the individual dietary counseling.

DETAILED DESCRIPTION:
The investigators will investigate the tastes (umami, bitter, salty, sweet and sour) that the patients prefers in order to increase the energy intake and reduce the risk of weight loss and loss of fat-free mass for patients with hematological cancer.

The study will be conducted as a single blinded randomized controlled trial. 40 patients will be recruited, and will be divided into two groups; the intervention group and the control group. The patients will not know which group they belong to.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Able to understand the "Participant Information" paper
* Diagnosed with hematological cancer
* Must be undergoing chemotherapy (at least one treatment during the study)
* Outpatient
* Be able to take pictures of meals (and send to the sub-investigators)
* Be able to speak and read the danish language

Exclusion Criteria:

* Pacemaker

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-03-28 (Actual); Primary Completion 2022-07-28 (Estimated); Study Completion 2022-08-15 (Estimated)

PRIMARY OUTCOMES:
Consumption of energy as a percentage of estimated need | 6 weeks
  difference - before and after intervention

SECONDARY OUTCOMES:
Fat-free-mass and fat-mass in percent (bioimpedance measurement) | 6 weeks
  difference - before and after intervention
Satisfaction (measured with EROTC QLQ-C30 version 3.0) | 6 weeks
  difference - before and after intervention. Higher scores means worse outcome. Lower scores means better outcomes.
Hand-grip-strength (measured with a dynamometer) | 6 weeks
  difference - before and after intervention
Body weight | 6 weeks
  difference - before and after intervention
Protein intake | 6 weeks
  difference - before and after intervention
Burning/pain in the mouth (measured on a scale) | 6 weeks
  difference - before and after intervention measured with Likert scale (1 to 5). Higher scores means a worse outcome. Lower scores means better outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Hematology, Roskilde, Denmark

IPD SHARING:
Plan to Share IPD: No